CLINICAL TRIAL: NCT06555653
Title: The Effect of Video-based Multimedia Information Before Amniocentesis on Pain, Anxiety and Pregnancy Outcomes
Status: Completed | Type: Observational
Sponsor: Başakşehir Çam & Sakura City Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2023-571
Record Dates: First submitted 2024-08-02; First posted 2024-08-15 (Actual); Last update posted 2024-08-15 (Actual); Status verified 2024-08

CONDITIONS: Amniocentesis; Video Information
Keywords: Video-based information, amniocentesis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Subjects received video-based multmedia information
  Interventions: Other: Video based multimedia information
- Subjects received traditional written information

INTERVENTIONS:
Other: Video based multimedia information — The intervention group was shown a 5 minute informational video before amniocentesis including definition of amniocentesis, its indications, the setup of amniocentesis room, the purpose and steps of the procedure, potential complications and how to manage them
  Groups: Subjects received video-based multmedia information

SUMMARY:
The goal of this clinical trial is to assess the effect of video-based multimedia information before amniocentesis on pain, anxiety and pregnancy outcomes

DETAILED DESCRIPTION:
Amniocentesis is the most commonly used invasive prenatal diagnostic test. This study aimed to investigate the effect of video-based multimedia information (MMI) on the anxiety and pain levels of patients undergoing amniocentesis.

All consecutive women aged 18-45 years scheduled for amniocentesis were included in this prospective randomized controlled study. Subjects were assigned to receive video-based MMI or traditional written information (controls). Anxiety levels were assessed at the first admission using the State and Trait Anxiety Inventory-State (STAI-S). After MMI and written information, STAI-S was repeated before the procedure. A standard amniocentesis procedure was performed on all patients by the same perinatology physicians. After amniocentesis, a Likert scale was used to evaluate the ease of the procedure and patient satisfaction, and a visual analog scale was used to evaluate pain. Pregnancy results and amniocentesis results were noted

ELIGIBILITY:
Inclusion Criteria:

* All consecutive women aged 18-45 years scheduled for amniocentesis

Exclusion Criteria:

-

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — All consecutive women aged 18-45 years scheduled for amniocentesis
Study Population: Women who received video based multimedia information about amniocentesis
Sampling Method: Probability Sample
Enrollment: 160 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2024-06-20 (Actual)

PRIMARY OUTCOMES:
To assess the effect of video based information on pain levels | 01.12.2023- 01.04.2024
  Subjects were assigned to receive video-based MMI or traditional written information (controls). A standard amniocentesis procedure was performed on all patients by the same perinatology physicians. After amniocentesis a visual analog scale was used to evaluate pain.
To assess the effect of video based information on anxiety | 01.12.2023- 01.04.2024
  Subjects were assigned to receive video-based MMI or traditional written information (controls). Anxiety levels were assessed at the first admission using the State and Trait Anxiety Inventory-State (STAI-S). After MMI and written information, STAI-S was repeated before the procedure.
To assess the effect of video based information on ease of procedure | 01.12.2023- 01.04.2024
  Subjects were assigned to receive video-based MMI or traditional written information (controls). A standard amniocentesis procedure was performed on all patients by the same perinatology physicians. After amniocentesis, a Likert scale was used to evaluate the ease of the procedure and patient satisfaction,
To assess the effect of video based information on pregnancy outcome | 01.12.2023- 01.04.2024
  Subjects were assigned to receive video-based MMI or traditional written information (controls).The birth outcomes were compared between the two groups in terms of live birth, termination of pregnancy, and intrauterine death.

CONTACTS AND LOCATIONS:
Overall Officials: Nihal Callıoglu, Study Director — Başakşehir Çam & Sakura City Hospital
Locations (1):
- Basaksehir Cam and Sakura City Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No